CLINICAL TRIAL: NCT01910259
Title: A Multi-arm Phase IIB Randomised, Double Blind Placebo-controlled Clinical Trial Comparing the Efficacy of Three Neuroprotective Drugs in Secondary Progressive Multiple Sclerosis.
Brief Title: MS-SMART: Multiple Sclerosis-Secondary Progressive Multi-Arm Randomisation Trial
Acronym: MS-SMART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government); National Institute for Health Research, United Kingdom (Other Government); National Multiple Sclerosis Society (Other); University of Edinburgh (Other); Queen Mary University of London (Other); Keele University (Other); University of Sheffield (Other); University of Leeds (Other); University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12/0219
Record Dates: First submitted 2013-07-19; First posted 2013-07-29 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: Secondary Progressive Multiple Sclerosis; Neuroprotective; Repurposed drugs; Brain atrophy; Percentage Brain Volume Change; Magnetic Resonance Imaging; Optical Coherence Tomography; Cerebrospinal fluid; Amiloride; Riluzole; Double blind; Placebo; Fluoxetine
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Amiloride; Riluzole; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Amiloride (Experimental): Amiloride 5 mg twice per day (5 mg once per day for first 4 weeks) for 96 weeks
  Interventions: Drug: Amiloride
- Riluzole (Experimental): Riluzole 50 mg twice per day (50 mg once per day for first 4 weeks) for 96 weeks
  Interventions: Drug: Riluzole
- Fluoxetine (Experimental): Fluoxetine 20 mg twice per day (20 mg once per day for first 4 weeks) for 96 weeks
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Matched placebo 1 capsule twice per day (1 capsule a day for first 4 weeks) for 96 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amiloride — Comparison with placebo
  Arms: Amiloride
Drug: Riluzole — Comparison with placebo
  Arms: Riluzole
Drug: Fluoxetine — Comparison with placebo
  Arms: Fluoxetine
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
Multiple sclerosis (MS) is a disabling and progressive neurological disease that affects approximately 100,000 people in the UK. Many patients with MS experience two phases of disease; early MS (also called relapsing remitting MS, RRMS) and late MS (also called secondary progressive MS (SPMS). Early MS is due to inflammation of the nerves and the insulation (called myelin) that surrounds the nerves. Early MS is often characterised by periods of "attacks" interspersed with periods of "remission" with no or low disease symptoms. Late or progressive MS, which affects the majority of patients and typically emerges after 10-15 years of disease, results from actual nerve death (also called neurodegeneration). The progressive stage of disease results not in individual attacks but slow, cumulative and irreversible disability affecting walking, balance, vision, cognition, pain control, bladder and bowel function. Critically, and unlike early disease, there is no proven treatment for the late stage of MS. This is therefore an urgent and major unmet health need. MS-SMART directly addresses this need and will evaluate in this clinical trial three drugs (fluoxetine, riluzole or amiloride), all of which have shown some promise in MS, and in particular in SPMS. The trial is randomised and blinded. Randomisation means patients can get any one of the three active drugs or the inactive placebo/dummy; blinded means that neither patients nor the doctors will know which drug or placebo patients are receiving. Randomisation and blinding are standard approaches in clinical trials to ensure unbiased testing of drugs. All patients in MS-SMART will have periodic MRI (magnetic resonance imaging) brain scans and after 96 weeks these will be analysed. We will then compare the scans of each drug to the placebo or dummy to see if any of the drugs slow the rate of brain shrinkage that normally occurs in SPMS. This measured change in brain size is the primary (major) outcome of MS-SMART.

DETAILED DESCRIPTION:
MS-SMART will test the efficacy and mechanism of action of three repurposed drugs (fluoxetine, riluzole and amiloride). All three drugs are in human use and have a good safety record. Critically for the purpose of MS-SMART they all have shown promise in early phase human MS clinical trials and target one or more of the pivotal neurodegenerative causing pathways implicated in SPMS. This is a Type B trial, as the IMPs are all in human use, have a good safety profile but are not currently used for this patient population.

The major need for patients with established and progressive MS is neuroprotective or disease modifying treatments that will slow or even stop disease progression. This study will evaluate three highly promising putative neuroprotective drugs as well as comprehensively address several of the current knowledge gaps related to the understanding of neuroprotection and neurodegeneration in SPMS through MRI and CSF examination.

MS-SMART is a multicentre, multi-arm, double blind, placebo-controlled phase IIb randomised controlled trial. A total of 440 patients with SPMS, with an entry criteria of an EDSS score of 4.0-6.5 will be equally randomised to receive placebo or one of the three active agents (fluoxetine 20mg bd, amiloride 5mg bd or riluzole 50mg bd). Patients will be followed up for 96 weeks with outcome-data collected after 0, 24, 48 and 96 weeks. That is, the duration of the trial for a trial participant is 96 weeks (a telephone assessment at week 100, 4 weeks post completion will be conducted). This is standard practice for phase II trials in SPMS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SPMS. Steady progression rather than relapse must be the major cause of increasing disability in the preceding 2 years. Evidence of progression, either an increase of at least one point in EDSS or clinical documentation of increasing disability in patient notes
* Expanded Disability Status Scale (EDSS) 4.0-6.5
* Aged 25 to 65 inclusive
* Women and men with partners of childbearing potential must be using an appropriate method of contraception to avoid any unlikely teratogenic effects of the 3 drugs from time of consent, to 6 weeks after treatment inclusive
* Women must have a negative pregnancy test within 7 days prior to the baseline visit unless not of child bearing potential (e.g. have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy or they are postmenopausal)
* Willing and able to comply with the trial protocol (e.g. can tolerate MRI and fulfils the requirements for MRI, e.g. not fitted with pacemakers or permanent hearing aids), ability to understand and complete questionnaires
* Written informed consent provided

Exclusion Criteria:

* Pregnancy or breast feeding patients
* Baseline MRI scan not of adequate quality for analysis (e.g. too much movement artefact)
* Significant organ co-morbidity (e.g. malignancy or renal or hepatic failure)
* Relapse within 3 months of baseline visit
* Patients who have been treated with iv or oral steroids for an MS relapse/progression within 3 months of baseline visit (these patients can undergo future screening visits once the 3 month window has expired), patients on steroids for another medical condition may enter as long as the steroid prescription is not for multiple sclerosis (relapse/ progression).
* Use of Simvastatin at 80mg dose within 3 months of baseline visit (lower doses of Simvastatin and other statins are permissible)
* Commencement of fampridine within 6 months of baseline visit
* Use of immunosuppressants (e.g. azathioprine, methotrexate, cyclosporine) or disease modifying treatments (β-interferons, glatiramer) within 6 months of baseline visit
* Use of fingolimod/fumarate/teriflunomide/laquinomod/or other experimental disease modifying treatment (including research of an investigational medicinal product) within 12 months of baseline visit
* Use of mitoxantrone/ natalizumab/ alemtuzumab/ daclizumab if treated within 12 months of baseline visit
* Primary progressive MS
* Relapsing-remitting MS
* Known hypersensitivity to the active substances and their excipients to any of the active drugs for this trial
* Use of: lithium, chlorpropamide, triamterene and spironolactone within 6 months of the baseline visit
* Current use of potassium supplements
* Current use of tamoxifen
* Current use of herbal treatments containing St. John's Wort
* Significant signs of depression
* Use of an SSRI within 6 months of the baseline visit
* Use of monoamine oxidase inhibitors, phenytoin, L-tryptophan) and/or neuroleptic drugs within 6 months of the baseline visit
* A Beck Depression Index score of 19 or higher
* Bipolar disorder
* Receiving or previously received Electro-Convulsive Therapy
* Epilepsy/seizures
* Glaucoma
* Patients with a history of bleeding disorders or currently on anticoagulants Routine screening blood values (LFT) >/ 3 x upper limit of normal (ULN) of site reference ranges (ALT/AST, bilirubin,ˠGT) Potassium <2.8mmol/l or >5.5mmol/l
* Sodium <125mmol/l
* Creatinine >130μmol/l
* WBCs <3 x 109/l
* Lymphocytes <0.8 x 109/l
* Neutrophil count <1.0 x 109 /l
* Platelet count <90 x 109 /l
* Haemoglobin <80g/l

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
MRI-derived Percentage Brain Volume Change (PBVC). | 2 years
  To establish whether a drug, from a panel of 3 leading candidate neuroprotective drugs, slows the rate of brain volume loss in SPMS over 96 weeks using MRI-derived percentage brain volume change (PBVC).

SECONDARY OUTCOMES:
Multi-arm trial strategy assessment | 2 years
  To establish that a multi-arm trial strategy is an efficient way of screening drugs in SPMS and can become the template for future work.
Count of new and enlarging T2 lesions | 2 years
  To explore any anti-inflammatory drug activity using the count of new and enlarging T2 lesions.
Pseudo-atrophy | 6 months
  Examining for evidence of pseudo-atrophy (to ensure reliability of the primary outcome measure).
Clinical measure of neuroprotection | 2 years
  To examine the clinical effect of neuroprotection as measured by clinician - EDSS, MSFC, SDMT, SLCVA, relapse rate and patient reported outcome measures - MSIS29 v2, MSWS v2, Pain - NPRS and BPI and Fatigue - NFI.
Health economics | 2 years
  To collect basic health economic data (EQ-5D) to inform future phase III trials.

OTHER OUTCOMES:
New T1 hypotense lesion count | 2 years
  Persistent new T1 hypointense lesion count to assess neuroprotection in new lesions.
Grey matter volume change | 2 years
  Grey matter volume change to assess cortical neuroprotection.
MR spectroscopy measured N-acetyl aspartate, myoinositol and glutamate | 2 years
  MR spectroscopy (MRS) to measure N-acetyl aspartate (reversal of neuronal mitochondrial dysfunction), myoinositol (prevention of glial cell inflammation) and glutamate (prevention of excitotoxicity).
Myelination | 2 years
  Magnetic Transfer Ratio (MTR) to evaluate myelination.
Cervical cord imaging | 2 years
  Cervical cord imaging to assess cord neuroprotection.
Composite MRI/disability scores | 2 years
  Composite MRI/disability scores to increase sensitivity and study interaction of treatment mechanisms.
Cerebrospinal fluid (CSF) neurofilament levels | 2 years
  Quantification of Cerebrospinal fluid (CSF) neurofilament levels to measure neuroprotection.
Optical Coherence Tomography (OCT) measured Retinal Nerve Fibre Layer (RNFL) thickness | 2 years
  Optical Coherence Tomography (OCT) measured Retinal Nerve Fibre Layer (RNFL) thickness as a measure of neuroprotection.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Chataway, Principal Investigator — University College, London; Siddharthan Chandran, Principal Investigator — University of Edinburgh
Locations (13):
- United Kingdom (13):
  - Anne Rowling Regenerative Neurology Clinic, Royal Infirmary of Edinburgh, Edinburgh
  - Gartnavel Royal Hospital, 1055 Great Western Road, Glasgow
  - Brighton and Sussex University Hospitals, Haywards Heath
  - St James's University Hospital, Leeds
  - The Walton Centre, Liverpool
  - The National hospital for Neurology and Neurosurgery, University College London, London
  - The Royal Victoria Infirmary, Newcastle
  - Queens Medical Centre, Nottingham
  - John Radcliffe Hospital, Oxford University Hospitals NHS Trust, Oxford
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield
  - University Hospital of North Staffordshire, Stoke-on-Trent
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] John N, Li Y, De Angelis F, Stutters J, Prados Carrasco F, Eshaghi A, Doshi A, Calvi A, Williams T, Plantone D, Phan T, Barkhof F, Chataway J; MS-SMART Investigators; Ourselin S, Braisher M, Beyene T, Bassan V, Zapata A, Chandran S, Connick P, Lyle D, Cameron J, Mollison D, Colville S, Dhillon B, Ross M, Cranswick G, Walker A, Smith L, Giovannoni G, Gnanapavan S, Nicholas R, Rashid W, Aram J, Ford H, Pavitt SH, Overell J, Young C, Arndt H, Duddy M, Guadagno J, Evangelou N, Craner M, Palace J, Hobart J, Sharrack B, Paling D, Hawkins C, Kalra S, McLean B, Stallard N, Bastow R. Brain reserve and physical disability in secondary progressive multiple sclerosis. BMJ Neurol Open. 2024 Sep 7;6(2):e000670. doi: 10.1136/bmjno-2024-000670. eCollection 2024. PMID 39262426
- [Derived] Williams T, Alexander S, Blackstone J, De Angelis F, John N, Doshi A, Beveridge J, Braisher M, Gray E, Chataway J; MS-SMART and MS-STAT2 Investigators. Optimising recruitment in clinical trials for progressive multiple sclerosis: observational analysis from the MS-SMART and MS-STAT2 randomised controlled trials. Trials. 2022 Aug 9;23(1):644. doi: 10.1186/s13063-022-06588-z. PMID 35945550
- [Derived] Chataway J, De Angelis F, Connick P, Parker RA, Plantone D, Doshi A, John N, Stutters J, MacManus D, Prados Carrasco F, Barkhof F, Ourselin S, Braisher M, Ross M, Cranswick G, Pavitt SH, Giovannoni G, Gandini Wheeler-Kingshott CA, Hawkins C, Sharrack B, Bastow R, Weir CJ, Stallard N, Chandran S; MS-SMART Investigators. Efficacy of three neuroprotective drugs in secondary progressive multiple sclerosis (MS-SMART): a phase 2b, multiarm, double-blind, randomised placebo-controlled trial. Lancet Neurol. 2020 Mar;19(3):214-225. doi: 10.1016/S1474-4422(19)30485-5. Epub 2020 Jan 22. PMID 31981516
- [Derived] Connick P, De Angelis F, Parker RA, Plantone D, Doshi A, John N, Stutters J, MacManus D, Prados Carrasco F, Barkhof F, Ourselin S, Braisher M, Ross M, Cranswick G, Pavitt SH, Giovannoni G, Gandini Wheeler-Kingshott CA, Hawkins C, Sharrack B, Bastow R, Weir CJ, Stallard N, Chandran S, Chataway J; UK Multiple Sclerosis Society Clinical Trials Network. Multiple Sclerosis-Secondary Progressive Multi-Arm Randomisation Trial (MS-SMART): a multiarm phase IIb randomised, double-blind, placebo-controlled clinical trial comparing the efficacy of three neuroprotective drugs in secondary progressive multiple sclerosis. BMJ Open. 2018 Aug 30;8(8):e021944. doi: 10.1136/bmjopen-2018-021944. PMID 30166303
- See also: Trial website — http://ms-smart.org